CLINICAL TRIAL: NCT04087499
Title: Potential Role of Acupuncture Treatment in Neuronal and Network Dysfunction in Patients With Vascular Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201802103A3
Record Dates: First submitted 2019-08-18; First posted 2019-09-12 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-08

CONDITIONS: Vascular Cognitive Impairment
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regular medication treatment (Sham Comparator): regular medication treatment
  Interventions: Device: Acupuncture
- acupuncture and regular medication treatment (Experimental): acupuncture and regular medication treatment
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — acupuncture treatment on selected acupoint

SUMMARY:
Vascular cognitive impairment (VCI) is a broad dimensional term, ranging from mild cognitive impairment without incapacity on activity of daily living to vascular dementia (VaD), referred to as significant cognitive impairment and decline in function status.

In this three-year project, we aim to evaluate the effects of biochemical data, early clinical variables, neuroimaging results, and intervention of acupuncture treatment on vascular event related cognitive impairment in crossectional analysis and longitudinal follow-up.

DETAILED DESCRIPTION:
Stroke is a common cerebrovascular disease of the central nervous system leading to serious medical complication. It results in a high mortality rate and increased disability rate. Stroke survivors may have long-lasting consequences, including motor dysfunction, sensibility dysfunction, and cognitive impairment]. Cognition is a key component of rehabilitation and recovery; therefore it is associated with poor engagement in rehabilitee and outcomes including increased mortality. As vascular dementia (VaD) is considered the second-most-common type of dementing illness, accounting for a significant proportion of total dementia case, vascular cognitive impairment (VCI) is a broader dimensional term, ranging from mild cognitive impairment without incapacity on activity of daily living to VaD, referred to as significant cognitive impairment and decline in function status.

Acupuncture is an ancient Chinese medical technique in which fine, stainless steel needles are inserted into certain anatomical locations of the body surface to elicit neurohormonal responses of the body system via nerve stimulation. Acupuncture are reported to be probably effective in improving cognitive function in vascular dementia animal models via multiple mechanisms such as anti-apoptosis, antioxidative stress reaction, and metabolism enhancing of glucose and oxygen.

Motor features may not parallel to the cognitive changes, it will serve as the disease progression marker. Unified Parkinson's Disease Rating Scale (UPDRS)-part III scores and NIH Stroke Scale (NIHSS) will be used.

1. At Kaohsiung Chang Gung Memorial Hospital, all the patients (n=80) will be included and receive a Standardized Acupuncture intervention; 40 will be treated with regular medication; 40 will be treated with acupuncture and regular medication.
2. For acupressure program, all participants are treated in supine position, and a certified TCM physician applied firm pressure (3 to 5 kg of pressure) with fingertips in a circular motion at a speed of 2 circles per second for a duration of one minute per acupoint. The complete process lasts for 8 minutes.

Cognitive function, Motor function, Mood and Sleep will be evaluated at baseline and follow-up period of time at 3 month, 6 month, and 12 month.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the diagnostic criteria of vascular cognitive impairment

Exclusion Criteria:

1. Systemic inflammatory disease with on-going treatment
2. Severe psychiatric disease, such as major depressive disorder or schizophrenia
3. Severe traumatic brain injury
4. Unable to tolerate exam of brain MRI

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline sleep quality at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Analogous variables were extracted from actigraphy. The sleep variables collected were sleep start time, sleep end time, sleep duration, sleep efficiency, and wake after sleep onset time, and the activity variables collected were heart rate activity score,activity amount, and activity intensity

SECONDARY OUTCOMES:
Change from baseline neuro-behavioral performances at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Cognitive Abilities Screening Instrument (CASI). In addition to general cognitive performance, CASI was used to evaluate specific domains, including short-term memory, attention and concentration, abstraction, visual construction, language, and list-generating fluency.
Change from baseline motor function (UPDRS) at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Unified Parkinson's Disease Rating Scale (UPDRS)-part III scores for parkinsonian features.
Change from baseline motor function (NIHSS) at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  NIH Stroke Scale (NIHSS) score 0-24.
Change from baseline continuous motor function at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Physical activity was measured using accelerometers.
Change from baseline memory performances at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Verbal memory were evaluated by using Chinese Version Verbal Learning Test (CVVLT).Visual-spatial abilities.
Change from baseline executive performances at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Attention and executive function was evaluated by Trail Making Test B.
Change from baseline executive performances (Stroop interference test) at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Attention and executive function was evaluated by Stroop interference test.
Change from baseline executive performances (calculation) at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  As the calculation ability depends on executive function, calculation ability was evaluated to reflect part of executive function.
Change from baseline abstract thinking at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Abstract reasoning was evaluated by using similarities (conceptualization) in frontal assessment battery-Similarities.
Change from baseline language performances at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Boston Naming Test were used to evaluate language ability in naming.
Change from baseline fluency performances at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  Semantic category fluency.
Change from baseline neuropsychiatric symptoms at 3 months, 6 months, 12 months | 3 months, 6 months, 12 months
  The neuropsychiatric symptoms of the participants were measured using the Neuropsychiatric Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: YaTing Chang, MD,PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No